CLINICAL TRIAL: NCT06670976
Title: Pilot Study of Soft Tissue Sarcoma Treated With Propranolol and Radiation
Brief Title: Propranolol Plus Standard Radiation Therapy Before Surgery for the Treatment of Patients With Soft Tissue Sarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: to be submitted at a later date
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3905123; NCI-2024-08858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3905123 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Propranolol; Radiotherapy; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (propranolol, RT, surgery) (Experimental): Patients receive propranolol PO BID for 2 weeks prior to standard of care RT (weeks 1 and 2) and then during and after standard of care RT (weeks 3-7). Treatment continues in the absence of disease progression or unacceptable toxicity until the time of standard of care surgery (week 8). Additionally, patients undergo PET scan and/or CT scan during screening and may undergo blood and tissue biopsy sample collection throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Drug: Propranolol; Radiation: Radiation Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy sample collection
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Propranolol — Given PO
  Other Names: 1-[(1-Methylethyl)amino]-3-(1-naphthalenyloxy)-2-propanol
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I trial tests the safety, tolerability and impact of adding propranolol to standard radiation therapy (RT) before surgery for the treatment of patients with soft tissue sarcoma. Sarcomas are a diverse group of rare tumors arising from connective tissue. Approximately 13,000-16,000 new cases of sarcomas arise in the United States annually. Sarcoma management involves multidisciplinary team decision making and treatment is multimodal utilizing chemotherapy (if needed) and RT prior to surgical intervention. Propranolol is a drug that has been used for many years for high blood pressure by blocking both beta-1 and beta-2 adrenergic receptors. Preclinical data suggests that blocking the beta-2 adrenergic receptors can improve the response to both chemotherapy and radiation. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. RT before surgery makes the tumor smaller and reduces the amount of tissue that needs to be removed during surgery. Surgery is the most common treatment for soft tissue sarcoma. Giving propranolol with standard RT before surgery may be safe, tolerable and impactful in treating patients with soft tissue carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety and tolerability of adding propranolol to standard RT for soft tissue sarcoma.

SECONDARY OBJECTIVE:

I. To evaluate the response of tumor immune microenvironment to treatments for patients.

OUTLINE:

Patients receive propranolol orally (PO) twice daily (BID) for 2 weeks prior to standard of care RT (weeks 1 and 2) and then during and after standard of care RT (weeks 3-7). Treatment continues in the absence of disease progression or unacceptable toxicity until the time of standard of care surgery (week 8). Additionally, patients undergo positron emission tomography (PET) scan and/or computed tomography (CT) scan during screening and may undergo blood and tissue biopsy sample collection throughout the trial.

After completion of study treatment, patients are followed up at 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Eligible for curative-intent radiation therapy for a soft tissue extremity sarcoma
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known hypersensitivity to propranolol
* Contraindication to beta-blockers e.g.; uncontrolled depression, unstable angina pectoris, uncontrolled heart failure (New York Heart Association [NYHA] grade III or IV), hypotension (systolic blood pressure < 85 or fasting plasma glucose > 160 mg/dL at screening), symptomatic peripheral arterial disease or Raynaud's syndrome, untreated pheochromocytoma, current nondihydropyridines calcium channel blocker use (such as verapamil, diltiazem) or rhythm control agents such as digoxin and amiodarone. Patients with pacemakers will be excluded
* Patients cannot be on propranolol and another beta-blocker simultaneously. Patients already on beta-blockers can (with approval and under supervision of their primary care physician and/or cardiologist) may choose to stop their current beta-blocker and switch to propranolol for the duration of the study
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 5 weeks post-surgery
  Will evaluate safety and tolerability of adding propranolol to standard radiation therapy for soft tissue sarcoma. Will determine the occurrence of a grade 3 or higher treatment related adverse events. Will summarize using frequencies and relative frequencies, with the grade 3 or higher toxicity rate estimated using a 90% credible region obtained by Jeffrey's prior method. Will summarize toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) by attribution and grade using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Ribonucleic acid sequencing | Up to 12 weeks
  Will evaluate with biopsy specimens. Will summarize using the mean and standard deviation, and graphically using line and mean plots. Will be modeled as a function of time and a random patient effect using linear mixed models. Tests about the appropriate contrast of model estimates will be used to evaluate changes over time. All model assumptions will be verified graphically and transformations applied as appropriate.
Changes in immune markers | Up to 12 weeks
  Changes in immune markers of CD8+ and CD4+ T cells and polymorphonuclear-myeloid-derived suppressor cells will be determined by flow cytometry in peripheral blood. Will summarize using the mean and standard deviation, and graphically using line and mean plots. Will be modeled as a function of time and a random patient effect using linear mixed models. Tests about the appropriate contrast of model estimates will be used to evaluate changes over time. All model assumptions will be verified graphically and transformations applied as appropriate.
Catecholamines | Up to 12 weeks
  Will correlate the levels of catecholamines and metabolites in peripheral blood. Will summarize using the mean and standard deviation, and graphically using line and mean plots. Will be modeled as a function of time and a random patient effect using linear mixed models. Tests about the appropriate contrast of model estimates will be used to evaluate changes over time. All model assumptions will be verified graphically and transformations applied as appropriate.
Metabolites | Up to 12 weeks
  Will correlate the levels of catecholamines and metabolites in peripheral blood. Will summarize using the mean and standard deviation, and graphically using line and mean plots. Will be modeled as a function of time and a random patient effect using linear mixed models. Tests about the appropriate contrast of model estimates will be used to evaluate changes over time. All model assumptions will be verified graphically and transformations applied as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States